CLINICAL TRIAL: NCT01593423
Title: Integration of Small-scale Aquaculture With Homestead Food Production for Improved Household Food Security and Nutrition in Rural Cambodia
Brief Title: Food Security and Nutrition in Rural Cambodia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Tim Green, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H12-00451
Record Dates: First submitted 2012-04-20; First posted 2012-05-08 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2016-11

CONDITIONS: Household Food Security

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Homestead Food Production plus small pond aquaculture (Experimental)
  Interventions: Behavioral: Homestead Food Production plus small pond aquaculture
- plant-based Homestead Food Production (Active Comparator)
  Interventions: Behavioral: plant-based Homestead Food Production
- Control (Sham Comparator)
  Interventions: Behavioral: a comparison group

INTERVENTIONS:
Behavioral: plant-based Homestead Food Production — The village model farm will be provided with the necessary inputs to establish their farm including saplings seeds etc.
  Arms: plant-based Homestead Food Production
Behavioral: Homestead Food Production plus small pond aquaculture — In the case of the aquaculture arm a pond will be dug if there is not an existing pond and fingerlings and brood stocks will be provided. Hatcheries will be established if there is not one within a reasonable distance of the farms.
  Arms: Homestead Food Production plus small pond aquaculture
Behavioral: a comparison group — No intervention.
  Arms: Control

SUMMARY:
The project is a three arm randomized control trial in rural Cambodia designed to evaluate the impact of homestead food production (home gardens) with and without fish ponds versus control on household food security, dietary intake of women and youngest child, biochemical nutritional status of women, and household livelihoods over a 22 month period. Baseline and end line surveys will be conducted that involve questionnaires and a blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Must be represented by a woman.
* Must fall within the "poor" category in terms of community wealth rankings.
* Must have access to land (including homestead) for agriculture cultivation.
* Must have sufficient access to labor to undertake the homestead production activities.
* Must have a keen interest in participating in this action.
* Must have a least one child less than five years of age (in 80% of the target households).
* Have suitable land for pond and preferably own a small pond

In addition village model farm owners will:

* Have at least 1,200 square meters of land that can be used to establish the model farm;
* Have some disposable income to invest in the model farm for fencing and land preparation;
* Be productive, open to new ideas and willing to provide assistance to other households in the village;
* Be able and willing to maintain the VMF throughout the year;
* Commit to providing inputs and marketing support to group members at least during the project.

Exclusion Criteria:

* None, only that they don't meet the inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in nutritionally related biochemical measures at 22 months | At baseline and 22 months
  Haemoglobin (g/l) Haematocrit (%) Serum Ferritin (ng/ml) White Cell Count (x109/l) Red Cell Count (x1012/l) Mean Corpuscular Volume (fl) Mean Cell Haemoglobin (pg) Red Cell Width % Platelet Count (x109/l) Neutrophils % Eosinophils % Lymphocytes % Monocytes % Neutrophils # (x109/l) Eosinophils # (x109/l) Lymphocytes # (x109/l) Monocytes # (x109/l) C-Reactive Protein (mg/l)

SECONDARY OUTCOMES:
24-hour dietary recall | At baseline and 22 months
Mid-upper arm circumference | At baseline and 22 months
Household Food Security Scale | At baseline and 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Tim Green, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Rural Cambodia, Phnom Penh, Prey Veng, Cambodia

REFERENCES:
- [Derived] Williams BA, Cochrane KM, Fischer JAJ, Aljaadi AM, McAnena L, Ward M, McNulty H, Kroeun H, Green TJ, Whitfield KC, Karakochuk CD. The Homozygous Hemoglobin EE Variant Is Associated with Poorer Riboflavin Status in Cambodian Women of Reproductive Age. J Nutr. 2020 Jul 1;150(7):1943-1950. doi: 10.1093/jn/nxaa119. PMID 32433728
- [Derived] Michaux KD, Hou K, Karakochuk CD, Whitfield KC, Ly S, Verbowski V, Stormer A, Porter K, Li KH, Houghton LA, Lynd LD, Talukder A, McLean J, Green TJ. Effect of enhanced homestead food production on anaemia among Cambodian women and children: A cluster randomized controlled trial. Matern Child Nutr. 2019 May;15 Suppl 3(Suppl 3):e12757. doi: 10.1111/mcn.12757. PMID 31148398